CLINICAL TRIAL: NCT01708655
Title: Evaluation of the Accuracy and Reliability of B-Adrenergic Sweat Secretion Using an Evaporimeter to Assess CFTR Function in Cystic Fibrosis
Brief Title: Sweat Evaporimeter Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-1463
Record Dates: First submitted 2012-09-28; First posted 2012-10-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Sweat Evaporimeter
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sweat Evaporimeter measurement (Other): 1. 0.1 ml Carbachol, intraocular solution - diluted to 0.1 µg/ml in normal saline- dose 0.01 µg
  2. 0.2 ml Atropine sulphate, injection solution - diluted to 44 µg/ml in normal saline - dose 8.8 µg.
  3. 0.2 ml of the Beta cocktail injection solution diluted to 44 µg/ml atropine, 22 µg/ml isoproterenol and 4.6 mg/ml aminophylline in normal saline - dose:
     * 4.4 µg Isoproterenol hydrochloride, injection solution
     * 0.93 mg Aminophylline injection solution
     * 8.8 µg Atropine, injection solution
  Interventions: Other: Sweat Evaporimeter measurement

INTERVENTIONS:
Other: Sweat Evaporimeter measurement — 1. The forearm will be cleaned with distilled water. Mineral oil will be applied to the surface of the skin after each injection.
  2. intracutaneous injection of 0.2 ml of atropine
  3. Stimulation and inhibition of sweating in an adjoining "test" area. Assessment of sweat secretion with an evaporimeter for 10 minutes after:
     1. Intracutaneous injection of 0.1 ml carbachol for stimulation of the cholinergic sweat secretion.
     2. intracutaneous injection of 0.2 ml atropine to Inhibit cholinergic sweat secretion
     3. intracutaneous injection of 0.2 ml beta-cocktail (atropine isoproterenol and aminophylline) for stimulation of beta-adrenergic sweat secretion .
  The procedure would take about 45 minutes.

SUMMARY:
The investigators hypothesize that measurement of beta adrenergic induced sweat rate using an evaporimeter can accurately and reliably determine different levels of CFTR dysfunction within a spectrum of patients expressing various degrees of cystic fibrosis disease.

The investigators overall goal is to determine whether the evaporimeter technique of measuring beta-adrenergic induced sweat rate is capable of accurately and reliably identifying different levels of CFTR dysfunction, as a prerequisite before advancing this technique as biomarker assay into clinical trials.

DETAILED DESCRIPTION:
Preliminary data show that following β-adrenergic stimulation, evaporimetry can reliably measure sweat secretion that is: highly reproducible in healthy controls; reduced by 50% in CF obligate heterozygotes; and absent in CF patients carrying severe mutations on both alleles. Further, test- retest experiments suggest good intra-individual reliability. All these features satisfy the required criteria for a biomarker assay that is capable of assessing small increments in CFTR function in vivo in clinical trials designed to assess the effectiveness of correctors and potentiators of CFTR channel activity. Therefore, to provide additional evidence of the value of this novel technique the investigators will determine the accuracy and reliability of evaporimetry to measure Beta-adrenergic induced sweating in subjects with a range of CFTR channel activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 years and older.
2. Subject with or without confirmed diagnosis of CF.
3. Written informed consent obtained from subject.

Exclusion Criteria:

1. Patients who are participating in clinical trials evaluating the safety, efficacy or clinical outcome of drugs that may alter the CFTR Cl channel function will be excluded.
2. Any subject with a known hypersensitivity to any agonist used in the study or subjects receiving any drug (e.g. theophylline, antihypertensive agent) that might interfere with the investigations.
3. Subjects with active dermatitis or other chronic skin condition such as psoriasis or a strong allergic history.
4. Patients with a history of cardiac disease (including arrhythmias or hypertrophic obstructive cardiomyopathy).
5. CF patients with severe malnutrition (BMI<18 kg/m2).
6. CF patients with severe lung disease (FEV1<25%).
7. Subject who has been treated for pulmonary exacerbation or other acute illness within one week of the study procedure.
8. Any medical condition that, in the opinion of the investigator, will interfere with accurate conduct of the study.
9. Subjects who are pregnant or lactating.
10. Subject who is not able to stop inhalation therapy of β -adrenergic drugs 12 hrs before starting each test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Measurement of beta-adrenergic induced sweat rate using an evaporimeter can accurately and reliably determine different levels of CFTR dysfunction within a spectrum of patients expressing various degrees of CF disease. | Up to 2 hours
  The response patterns will be interpreted and classified by the study PI, as consistent or inconsistent to the published standards. The obtained measurements will be compared to the results obtained from a recently finished validation trial. According to the result of this trial the ranges were as followed: cholinergic response for all subjects 60±20 Evaporimeter units, beta-adrenergic response: Healthy control 51 ± 20 heterozygote -22 ±20, CF -1.4 ±2.

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Accurso, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States